CLINICAL TRIAL: NCT03886506
Title: Expanded Access to Provide Intramuscular Injections of PLX-PAD for the Treatment of Subjects With Critical Limb Ischemia (CLI) With Minor Tissue Loss Who Are Unsuitable for Revascularization
Brief Title: Expanded Access Treatment of Subjects With Critical Limb Ischemia (CLI) With Minor Tissue Loss Who Are Unsuitable for Revascularization
Status: No longer available | Type: Expanded Access
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PLX-CLI-05
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Biological: PLX-PAD — PLX-PAD 300×106 cells in a mixture containing 10% DMSO, 5% human serum albumin and Plasma-Lyte, will be administered via 30 IM injections (0.5 mL each) delivered into the leg twice,at 8 weeks interval.

SUMMARY:
A Phase III study of PLX-PAD for CLI patients with minor tissue loss who are unsuitable for revascularization has been initiated (PLX-CLI-03, PACE study). In parallel, this expanded access program (EAP) will be conducted to allow the treatment of patients who are ineligible to be enrolled in the PACE study.

The EAP treatment is administered in addition to standard of care of the subjects.PLX-PAD 300×106 cells in a mixture containing 10% DMSO, 5% human serum albumin and Plasma-Lyte, will be administered via 30 IM injections (0.5 mL each) delivered into the leg twice,at 8 weeks interval. The locations of injections of the PLX-PAD are detailed in Appendix 1.

Antihistamine treatment should be given at least 1 hour and no more than 1.5 hours prior to PLXPAD administration to ensure coverage for 24 hours, and as long as necessary post PLX-PAD treatment. Consider treatment with second generation H1 inhibitors such as Cetirizine 10 mg once per day.Subjects will be followed-up until 12 months after the 2nd treatment according to the schedule of routine medical visits at the medical institutions. In addition to this routine follow-up, a phone call will be made 12 months after 2nd treatment to inquire on the occurrence of subsequent intervention, amputation, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects between ages 45 to 99 years of age at the time of screening.
2. Subjects with a diagnosis of PAD due to atherosclerosis at the stage of CLI, with minor tissue loss up to the ankle level (ulcer/s and/or necrosis).
3. Ankle pressure (AP)≤70 mmHg or toe pressure (TP)≤ 50 mmHg in the index leg or transcutaneous oxygen pressure (TcPO2)≤ 30 mmHg.
4. Subject unsuitable for revascularization (by any method) in the index leg based on unfavorable risk-benefit assessment of the physician investigator. Unsuitability to revascularization should be based on any of the following:

   1. Anatomic considerations as: inappropriate target artery, diffuse/extensive tibial and/or peroneal artery lesions, inadequate distal run-off.
   2. Technical considerations as: inappropriate bypass conduit, failed recent revascularization.
   3. Medical considerations: subject's comorbidities.
5. Signed informed consent form.
6. Additionally, this protocol includes subjects who are not eligible for the ongoing phase III study with PLX-PAD in CLI (PLX-CLI-03) due to at least one of the following criteria:

   1. Evidence of active localized osteomyelitis secondary to contiguous focus of infection, unless amputation is expected within 1 months post PLX-PAD administration. In case of osteomyelitis, patients must be treated with antibiotics during screening and PLX-PAD administration or as long as there is evidence of active infection.
   2. Subject on renal replacement therapy or with eGFR <15 mL/min.
   3. Current treatment with high dose systemic steroids (prednisone equivalent >7.5 mg/day) or topical steroids on the index leg.
   4. History of autologous bone marrow transplantation (if not due to hematologic malignancy) or solid organ transplantation, clinically stable.
   5. Immunocompromised subjects due to disease for any reason, including immunosuppressive therapy, at screening (for steroid therapy, refer to the criterion c)
   6. CLI with major tissue loss (Rutherford Category 6) in the contralateral leg.
   7. Diabetes mellitus with glycosylated hemoglobin (HbA1c) >10% at Screening.
   8. HIV controlled by antiretroviral therapy
   9. Past drug or alcohol abuse.
   10. Known history of cancer is eligible if occurred beyond 2 years before screening.

Exclusion Criteria:

1. Non-atherosclerotic PAD and vasculitis (e.g., Buerger's disease [thromboangiitis obliterans], Takayasu's arteritis, etc.).
2. CLI with major tissue loss (Rutherford Category 6) in the index leg. Ulcers from venous or neuropathic origin if not associated with at least one ulcer from arterial origin.
3. Evidence of active infection in either leg (e.g., cellulitis, myositis) except localized osteomyelitis secondary to contiguous focus of infection, under antibiotic treatment.
4. Subject having undergone surgical/endovascular revascularization or major/minor amputation, in either leg, less than 1 month prior to Screening.
5. Planned or potential need for major/minor amputation or any revascularization of either leg within 1 month of EAP entry upon physician's judgment.
6. Aortoiliac stenosis or common femoral artery stenosis or otherwise suspicion of inadequate inflow to the index leg at the time of Screening.
7. Current evidence or sign supporting an assessment of life expectancy of less than 6 months.
8. Stroke or acute myocardial infarction within 3 months prior to Screening.
9. Severe congestive heart failure symptoms (New York Heart Association [NYHA] Stage IV) at screening.
10. Life-threatening ventricular arrhythmia - except in subjects with an implantable cardiac defibrillator at screening.
11. Uncontrolled severe hypertension during Screening.
12. Current or history of proliferative retinopathy.
13. Known active Hepatitis B virus or Hepatitis C virus infections at Screening. Pluristem, Ltd Expanded Access Protocol
14. Acquired immunodeficiency syndrome (AIDS), severe uncontrolled inflammatory disease,or severe uncontrolled autoimmune disease (e.g., ulcerative colitis, Crohn's disease, etc.).
15. Subjects at an increased risk of blood clotting or bleeding according to the Physician's judgment.
16. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3×ULN. Subjects with higher levels may be included if the condition associated with the increase in those liver enzymes is known and is considered clinically stable.
17. Current drug or alcohol abuse.
18. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending another investigational device or drug trial(s) unless in long-term follow-up phase (in which there is no IP administration).
19. Current use or use within 30 days prior to screening of wound dressing containing cells or growth factors like Apligraf®, or topical platelet derived growth factor.
20. Current use, planned use, or use within 15 days prior to treatment of hyperbaric oxygen therapy, spinal cord stimulation, or lumbar sympathectomy.
21. Exposure to allogeneic cell based therapy in the past or exposure to autologous cell therapy in the last 12 months before screening.
22. Known allergies to any of the following: dimethyl sulfoxide (DMSO), human serum albumin, bovine serum albumin.
23. History of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with intravenous steroids/epinephrine, known allergy to more than 3 allergens, or in the opinion of the Physician the subject is at high risk of developing severe allergic/hypersensitivity reactions.
24. History of severe atopic disease (including but not limited to chronic urticaria, respiratory allergy requiring oral steroids), or history of uncontrolled Asthma (Global Initiative for Asthma [GINA] III-IV).

    1. Pulmonary disease requiring supplemental oxygen treatment on a daily basis.
    2. History of acute transfusion reaction.
    3. History of allogeneic bone marrow transplantation.
    4. Active malignancy except for successfully resected skin basal cell carcinoma or not located on the index leg.
    5. Pregnant or lactation women
    6. Inability to understand and provide an informed consent.

Ages: 45 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - OBL-NJ Endovascular & Amputation Prevention, LLC,1429 Broad St., Clifton, NJ, Clifton, New Jersey
  - Holy Name Medical Center,718 Teaneck Road, Teaneck, New Jersey